CLINICAL TRIAL: NCT06195943
Title: Feasibility, Safety and Acceptability of a Mobile Health Delivered Exercise Training Program in Patients With Nonalcoholic Steatohepatitis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Milton S. Hershey Medical Center (Other)
Responsible Party: Principal Investigator, Justin Tondt, Assistant Professor of Family and Community Medicine and Public Health Sciences, Milton S. Hershey Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 22771
Record Dates: First submitted 2023-12-15; First posted 2024-01-08 (Actual); Last update posted 2025-07-29 (Actual); Status verified 2025-07

CONDITIONS: NASH - Nonalcoholic Steatohepatitis; NASH; Exercise; Liver
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Application Useage Arm (Other): Along with wearing their Fitbit daily, subjects will be asked to use El-Fit app to participant in daily exercise as much or a little as they want over the course of the study.
  Interventions: Behavioral: Exercise Intervention with use of El-Fit App

INTERVENTIONS:
Behavioral: Exercise Intervention with use of El-Fit App — Along with wearing their Fitbit daily, subjects will be asked to use El-Fit app to participant in daily exercise as much or a little as they want over the course of the study.

SUMMARY:
This study will be a pilot study to evaluate the feasibility, safety and acceptability of Exercise and Liver FITness (EL-FIT), a mHealth exercise training program previously validated in patients with cirrhosis in patients with nonalcoholic steatohepatitis.

ELIGIBILITY:
Inclusion Criteria:

* Adults age >18 years
* Evidence of NASH indicated by at least one of the following

  * Liver biopsy with evidence of steatohepatitis (NAS >=4) within 6 months of the screening interval or;
  * Historical Imaging study (e.g., ultrasound, CT, MRI) with hepatic steatosis and one of the following non-invasive tests within 6 months of the screening interval: i. FIB-4 >= 1.3 or; ii. NFS >= -1.44 or; iii. ELF >= 7.7 or; iv. VCTE kPa >=8 or; v. ARFI >=1.3 or; vi. FAST >= 0.35 or; vii. MRE kPa >=2.55 or; viii. MAST > 0.165 or;
* Possession of a smartphone

Exclusion Criteria:

* Active cardiac symptoms precluding participation in vigorous exercise
* Active or recent participation in exercise training program within the last 90 days
* Active or recent weight-loss supplement use within the last 90 days (does not include GLP-1 receptor agonist use)
* Active illicit substance use
* Cancer that is active
* Cirrhosis
* Exercise identified to be unsafe by study PI or EL-FIT mHealth program
* Inability to provide informed consent
* Inability to walk > 2 blocks
* Institutionalized/prisoner
* Other chronic liver disease (e.g., viral hepatitis)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-02-01 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Number of subjects that complete at least 50% of the exercise sessions | 8 weeks
  The primary study endpoint is feasibility of the use of the application, which is defined as >50% of subjects adhering to the exercise prescribed, defined as completing >50% of the sessions.

CONTACTS AND LOCATIONS:
Overall Officials: Justin G Tondt, MD, Principal Investigator — Penn State Health
Locations (1):
- Penn State Hershey Medical Center, Hershey, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No